CLINICAL TRIAL: NCT06256926
Title: A Prospective, Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of Curcuvail® of K Patel Phyto Extractions Pvt. Ltd. in Patients With Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: A Clinical Study of Curcuvail® in Patients With Non-alcoholic Fatty Liver Disease
Acronym: NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: COD Research Private Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSI2003; CSI2003, Version 2.0 (Other: K Patel Phyto Extractions Pvt. Ltd.)
Record Dates: First submitted 2021-12-08; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Fatty Liver Without Mention of Alcohol
MeSH Terms: interventions — Diarylheptanoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Product (Active Comparator): Test Product: Curcuvail® 250 mg capsule
  Interventions: Drug: Test Product: Curcuvail® 250mg capsule (Curcuma longa Extractcontaining 35% Curcuminoids)
- Placebo Product (Placebo Comparator): Placebo Product
  Interventions: Drug: Placebo product

INTERVENTIONS:
Drug: Test Product: Curcuvail® 250mg capsule (Curcuma longa Extractcontaining 35% Curcuminoids) — Curcuma longa Extract containing 35% Curcuminoids Dose: One capsule Frequency: Twice Daily Route of administration: Oral Duration of therapy: 60Days
  Other Names: Curcuvail® 250 mg capsule
  Arms: Drug Product
Drug: Placebo product — Placebo product Dose:One capsule Frequency: Twice Daily Route of administration: Oral Duration of therapy: 60Days
  Other Names: Placebo Comparator: Placebo Product
  Arms: Placebo Product

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease. It comprises a wide spectrum of disorders that range from simple steatosis to nonalcoholic steatohepatitis (NASH), advanced fibrosis, related cirrhosis, and even hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease. It comprises a wide spectrum of disorders that range from simple steatosis to nonalcoholic steatohepatitis (NASH), advanced fibrosis, related cirrhosis, and even hepatocellular carcinoma (HCC).

Currently there are no effective medications to cure NAFLD. Current treatments for NAFLD include weight reduction through lifestyle modification and exercise, insulin-sensitizing agents, lipid-lowering agents, and hepatoprotective drugs. However, the efficacy of these therapies is not satisfactory, some drugs may even induce liver toxicity. Thus, it is necessary to develop novel therapies that are effective and safe for the treatment of NAFLD.

Hence, K Patel Phyto Extractions Pvt. Ltd. has formulated Curcuvail®. Objective of the current study is to compare efficacy, safety and tolerability of test formulation Curcuvail® by administering the medications in the adult patients suffering from Non-alcoholic Fatty Liver Disease (NAFLD) and eligible to receive Curcuvail® as treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to any study-related activities being performed.
2. Able and willing to comply with the protocol, including availability for all scheduled study visits.
3. Male and Female patients aged between 18 years to 70, both inclusive.
4. Patients diagnosed with fatty liver (grades 1-3) based on liver ultrasonography.
5. Women of child bearing potential, (defined as women physiologically capable of becoming pregnant, unless they are using effective method of contraception during dosing of the investigational product) practicing any two acceptable methods of contraception.
6. Female patients with negative urine pregnancy test (only for female who has not completed 1 year after menopause & have not gone through hysterectomy or bilateral tubal ligation).

Exclusion Criteria:

1. Hypersensitivity to Curcuvail or related class of drugs or to any of the excipients of the formulation.
2. Fatty liver secondary to alcohol consumption.
3. History of regular alcohol consumption exceeding 14 drinks per week for female subjects or 21 drinks per week for male subjects (1 drink - 5 ounce [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within the previous 6 months from screening
4. Addicted Alcoholics and- or drug abusers.
5. History or presence of coronary, renal, pulmonary and thyroid disease.
6. AST and ALT more than 5 times ULN; Serum bilirubin more than ULN and Platelet Count less than 95,000 per microliter.
7. Patients using hypolipidemic medications as well as any drug known to affect hepatic function 4 weeks prior to randomization.
8. Difficulty in swallowing and retaining oral formulation.
9. Known HBs Ag positive, Anti HCV and HIV positive, hereditary defects of iron, copper and alpha- 1 antitrypsin deficient patients.
10. Hypothyroidism, obstructive sleep apnoea, total parenteral nutrition, short bowel syndrome, pancreatoduodenal resection which are secondary causes of NAFLD.
11. Patient has condition or is in a situation which, in the investigator's opinion, may have put the patient at a significant risk, may have confounded study results, or may have interfered significantly with the patient's participation in the study.
12. Participation in any other clinical study within 30 days before the first dose of Investigational Product.
13. Pregnant or Lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Change in NAFLD grading based on liver USG from baseline to day 60. | 60 Days
  NAFLD Grading:
  Grade 0: Lack of fat accumulation Grade 1: Mild Increase in echogenicity with normal visualization of the diaphragm and intra-hepatic vessel borders.
  Grade 2: Moderate increase in echogenicity with slightly impaired visualization of diaphragm and intra-hepatic vessel borders.
  Grade 3: Severe increase in echogenicity with markedly impaired visualization of diaphragm, intra-hepatic vessel borders, and posterior portion of the right hepatic lobe.

SECONDARY OUTCOMES:
AST to Platelet Ratio Index (APRI) | 60 Days
  APRI score assessed as change from baseline to day 60
Fibrosis score (kilopascals (kPa)) | 60 Days
  Fibrosis score evaluated by FibroScan and assessed as change from baseline to day 60
  Fibrosis score:
  F0 to F1 (No liver scarring or mild liver scarring): 2 to 7 kPa F2 (Moderate liver scarring) : 7.5 to 10 kPa F3 (Severe liver scarring) : 10 to 14 kPa F4 (Advanced liver scarring (cirrhosis)): 14 kPa or higher
Controlled Attenuation Parameter (CAP) score (decibels per meter (dB/m)) | 60 Days
  CAP score (dB/m) as evaluated by FibroScan and assessed as change from baseline to day 60.
Change in lipid profile from baseline to day 60 | 60 Days
  Change in lipid profile [total cholesterol, high density lipoprotein (HDL), low-density lipoprotein (LDL) and triglycerides represented as mg/dL] from baseline to day 60
Change in liver enzymes ALT and AST from baseline to day 60 | 60 Days
  Change in liver enzymes ALT (IU/L) and AST (IU/L) from baseline to day 60
Number (Frequency & percentage of patients) and type (severity and causality assessment) of AE (Adverse Event) and SAE (Serious Adverse Event). | Till 67 days from day of randomization
  AE (Adverse Event) and SAE (Serious Adverse Event) were evaluated during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mr. Nimesh Parekh, M.Sc., Study Director — Chief Operating Officer
Locations (1):
- Cod Research Pvt Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No